CLINICAL TRIAL: NCT06173453
Title: Factors Associated With Survival in Patients With a Positive Sample for Pneumocystis Jirovecii at the Strasbourg University Hospital: a Retrospective Study From 2016 to 2018
Brief Title: Factors Associated With Survival in Patients Having Pneumocystis Jirovecii
Acronym: JIROVECI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8722
Record Dates: First submitted 2023-06-15; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-06

CONDITIONS: Pneumocystis Jirovecii Infection
Keywords: P jirovecii Infection; Pneumocystis Infections; Pneumocystis jirovecii Infection; Pneumocystis jirovecii; Pneumonia; Pneumocystis
MeSH Terms: conditions — Pneumocystis Infections; Pneumonia; Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pneumocystis jirovecii is a fungus that can colonize the airways of some patients and be responsible for a disease called pneumocystosis in other patients and mainly in immunocompromised patients.

Pneumocystosis was mainly linked to HIV in the 1990s, but with the advent of new immunosuppressive molecules used in cancers or autoimmune diseases and with the increase in the number of transplants, the epidemiology has changed in recent years.

Studies on P. jirovecii-related mortality are only based on patients with pneumocystosis. As a result, patients who are simply colonized or patients who are sick but not treated are not taken into account in these studies. The investigators therefore wish to study the overall mortality at six weeks and at three months in all patients with a positive sample for P. jirovecii

ELIGIBILITY:
Inclusion criteria:

* Adult patients with a positive respiratory sample for P. jirovecii cared for in Strasbourg University Hospitals between 01/01/2016 and 31/12/2018. Positive samples are defined as a direct examination finding cysts or trophozoites after staining with May-Grunewald-Giemsa and/or Gomori-Grocott, a positive P. jirovecii PCR on sputum, tracheal aspirates or bronchial fluid -alveolar
* Subject not objecting to the reuse of their data for scientific research purposes.

Exclusion criteria:

- Subject having expressed its opposition to the reuse of its data for scientific research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a positive respiratory sample for P. jirovecii
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Survival at six weeks and three months after infection | six weeks after infection

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France